CLINICAL TRIAL: NCT06547567
Title: Promoting the Development of Autonomous Health Behaviors in Children and Adolescents Through Motivational Interviewing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PU IRB V1 (2023-10-31)
Record Dates: First submitted 2024-08-04; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing Group (Experimental): In addition to receiving the same health education intervention as the control group, the children and adolescents in the intervention group will undergo a group-based motivational interviewing intervention. This will be conducted by a professional team that has been trained and is qualified in motivational interviewing. The intervention will embody the spirit of motivational interviewing and the stages of group motivation development, primarily including: introductory tasks, exploratory tasks, expansion tasks, and action planning tasks.
  Interventions: Behavioral: Motivational Interviewing
- Health Education Intervention (No Intervention): Using various methods such as WeChat official accounts, video platforms, WeChat groups, and the distribution of health education pamphlets, we aim to disseminate scientific knowledge and practical skills related to healthy weight management and the prevention of overweight and obesity to children, adolescents, and their parents.

INTERVENTIONS:
Behavioral: Motivational Interviewing — In addition to receiving the same health education intervention as the control group, the children and adolescents in the intervention group will undergo a group-based motivational interviewing intervention. This will be conducted by a professional team that has been trained and is qualified in motivational interviewing. The intervention will embody the spirit of motivational interviewing and the stages of group motivation development, primarily including: introductory tasks, exploratory tasks, expansion tasks, and action planning tasks.
  Arms: Motivational Interviewing Group

SUMMARY:
1. Study Population

1. Sample Size: 150 children.
2. Randomization: This study will employ a randomized controlled intervention design. Participants will be stratified based on factors such as gender and age, and within each stratum, they will be randomly assigned in a 1:1 ratio to either the intervention group receiving motivational interviewing or the control group. The randomization process will be centralized and conducted by personnel not involved in the project.
3. Inclusion Criteria (all of the following must be met for inclusion):

   Both children/adolescents and their parents are willing to participate and demonstrate good compliance.

   Children/adolescents have a weight classified as normal, overweight, or obese. Age range: 10 to 14 years. Informed consent is obtained from both the child and the parent.
4. Exclusion Criteria (meeting any one of the following will result in exclusion):

Pathological obesity (e.g., due to endocrine disorders). Underweight. Clinically diagnosed severe mental illness or psychiatric disorders. Clinically diagnosed eating disorders (e.g., binge eating disorder). Physical developmental abnormalities or disabilities that prevent normal physical activity.

History of or plans to undergo pharmacological or surgical weight loss interventions within the next two years.

DETAILED DESCRIPTION:
Intervention Content Control Group: The control group will receive health education on weight management and the prevention of overweight and obesity through various channels, including WeChat official accounts, video platforms, WeChat groups, and the distribution of health education pamphlets. This aims to disseminate scientific knowledge and practical skills to children, adolescents, and their parents.

Intervention Group: In addition to receiving the same health education interventions as the control group, the intervention group will participate in group-based motivational interviewing. This will be conducted by a professional team that has been trained and certified in motivational interviewing techniques. The intervention will embody the principles of motivational interviewing and will follow a staged development approach, which includes:

Engagement tasks, exploration tasks, expansion tasks, action planning tasks.

Follow-up Survey This study will conduct a baseline survey and follow-up surveys at 3, 6, 12, 18, and 24 months post-intervention. The main survey indicators will include: personality traits, autonomous motivation, behavioral attitudes, subjective norms, perceived behavioral control, behavioral Intentions, stages of behavioral change, obesity-related behaviors, obesity status, mental health indicators.

ELIGIBILITY:
Inclusion Criteria:

* Both children/adolescents and their parents are willing to participate and demonstrate good compliance.
* Children/adolescents have a weight classified as normal, overweight, or obese.
* Age range: 10 to 14 years.
* Informed consent is obtained from both the child and the parent.

Exclusion Criteria:

* Pathological obesity (e.g., due to endocrine disorders).
* Clinically diagnosed severe mental illness or psychiatric disorders.
* Clinically diagnosed eating disorders (e.g., binge eating disorder).
* Physical developmental abnormalities or disabilities that prevent normal physical activity.
* History of or plans to undergo pharmacological or surgical weight loss interventions within the next two years.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Stages of Behavior Change | 2 years
  The main survey indicators include personality traits, autonomous motivation, behavioral attitudes, subjective norms, perceived behavioral control, behavioral intentions, stages of behavior change, obesity-related behaviors
Obesity Status (BMI) | 2 years
  The main survey indicators include obesity status, such as BMI